CLINICAL TRIAL: NCT06669286
Title: Retrospective Single Cohort Mono-center Study on Success and Safety of Navigated Implant Placement in Proximity of the Alveolar Nerve
Brief Title: Success and Safety of the Implant Placement Using Navigated Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Roberto Villa (Other)
Collaborators: Nobel Biocare Services AG (Unknown)
Responsible Party: Sponsor-Investigator, Roberto Villa, dentist, Clinica Odontoiatrica Villa
Organization: Clinica Odontoiatrica Villa (Other)
Other Study IDs: ClinicaOdontoiatricaVilla
Record Dates: First submitted 2024-10-26; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Edentulism
Keywords: navigated surgery; alveolar nerve; implant placement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: implant placement using navigated surgery near alveolar nerve — Dental implant placement in proximity of alveolar nerve (within 2 mm) using navigated surgery.

SUMMARY:
Subjects with severely atrophic mandibles were treated with implants and implant-based restorations. Subjects will be required to consent to study participation and data processing according to General Data Protection Regulation (GDPR). Implant positions were planned digitally in a dental software DTX Studio, and implants placed with navigated surgery (Nobel Biocare X-Guide). Implants eligible for this study must be placed 2 mm or less from the alveolar nerve. Implants placed are NobelParallel TiUnite and NobelActive TiUnite. All subjects were followed up for 1 year after surgery to monitor success and adverse events related to the alveolar nerve. Data analysis will include demographics, medical history, Cone-beam Computed Tomography (CBCT) scans/peri-apical x-ray data, soft tissue parameters, and adverse events.

DETAILED DESCRIPTION:
The study aims to evaluate the success and safety of immediate navigated implant placement in the atrophic mandible or post-extraction sockets near the alveolar nerve, as an alternative to guided bone regeneration followed by delayed implant placement.

This single-center retrospective study includes 20 subjects with severely atrophic mandibles or post-extraction sockets, followed for 1 year after implant placement.

The primary objective is to assess treatment success, defined as the implant supporting a dental prosthesis, no adverse events related to the alveolar nerve, and minimal bone loss around the implant. The secondary objective focuses on safety, particularly concerning the alveolar nerve. Subjects must meet specific inclusion criteria, such as implants placed within 2 mm of the alveolar nerve and being at least 18 years old and must have signed consent forms. Exclusion criteria include the absence of 1-year follow-up data.

Data collected includes demographic and medical history, plaque, bleeding, and gingival indices at pre-treatment and 1-year follow-up, and radiographic exams (CBCT and intra-oral radiographs) to assess bone levels. Written informed consent is required, and all data is de-identified and transferred to Switzerland for analysis, complying with EU regulations. This study aims to provide a less invasive alternative to traditional methods, potentially reducing the number of surgical interventions needed.

ELIGIBILITY:
Inclusion Criteria:

* Implants placed in 2 mm distance or less of the alveolar nerve
* Subject was at least 18 years old at the time of surgery
* Subject signed consent form
* Subject signed GDPR form

Exclusion Criteria:

* 1-year follow-up data on treatment success not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult subjects (18 years) treated at the investigator's private practice for severely atrophic sites or post-extraction sites (single tooth to max. 4 teeth) in the mandible with navigated surgery
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Treatment success after 1 year of implant placement | 1 year
  Treatment success is defined specific to this study as:
  * The implant supports a dental prosthesis
  * No adverse event related to the alveolar nerve
  * No or only minor bone loss around the implant

SECONDARY OUTCOMES:
Safety assessment with focus on alveolar nerve | 1 year
  The safety of the procedure will be evaluated based on the data collected from the adverse events and device deficiency issues. Based on the seriousness of the event it is categorized as either:
  * Adverse Event (AE)
  * Serious Adverse Event (SAE)• Adverse Device Effect (ADE) Serious Adverse Device Effect (SADE)
  * Unanticipated Serious Adverse Device Effect (USADE)
  * Device Deficiency (DD) Known issues associated with dental implant surgery include, but are not limited to, excessive bleeding during surgery, pain, alveolar wall fracture, partial or total anesthesia after surgery.

IPD SHARING:
Plan to Share IPD: Undecided